CLINICAL TRIAL: NCT03872011
Title: Initiation of Vitamin C, Thiamine and Hydrocortisone Therapy for Septic Shock in Adults: A Randomized Clinical Trial
Brief Title: Vitamin C, Thiamine and Hydrocortisone for the Treatment of Septic Shock
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Northern Jiangsu People's Hospital (Other)
Responsible Party: Principal Investigator, Qing-quan Lv, Principal Investigator, Northern Jiangsu People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019KY-145
Record Dates: First submitted 2019-03-04; First posted 2019-03-12 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Septic Shock
Keywords: septic shock; vitamin C; thiamine; hydrocortisone; mortality
MeSH Terms: conditions — Shock, Septic | interventions — Hydrocortisone; Ascorbic Acid; Thiamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin C,thiamine,hydrocortisone (Experimental): The combination of vitamin C, thiamine, hydrocortisone :
  Vitamin C 2g every 6 hours x 5-days Thiamine 200mg every 12 hours x 5-days Hydrocortisone 200mg as a continuous infusion x 5-days
  Interventions: Drug: Vitamin C,thiamine,hydrocortisone
- Placebo (Placebo Comparator): Normal Saline Solution (0.9%NaCl) in a volume to match all experimental arm components
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin C,thiamine,hydrocortisone — Vitamin C (2g) will be diluted in 100ml 0.9%NACL and administered ivd every 6 hours for 5 days or until participant is discharged from the ICU.
  Thiamine(200mg) will be diluted in 100ml 0.9%NACL and administered ivd every 12 hours for 5 days or until participant is discharged from the ICU. Hydrocortisone was administered 200 mg/d as a continuous infusion for 5 days or until participant is discharged from the ICU.
  Other Names: Ascorbic Acid; Vitamin B1
  Arms: Vitamin C,thiamine,hydrocortisone
Drug: Placebo — Normal saline (0.9% NaCl solution) volume to match all components
  Other Names: Normal saline
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether the combination therapy (vitamin C,thiamine and hydrocortisone) is effective in the treatment of septic shock.

DETAILED DESCRIPTION:
Septic Shock is a leading cause of morbidity and mortality in critically ill patients worldwide.

A potential benefit of vitamin C with thiamine and low-dose hydrocortisone in the treatment of septic shock has recently been described(PMID 27940189) . The patients with septic shock who received this combination of medications weaned off pressors earlier, suffered less organ failure, and had improved mortality. The doses of vitamin C used in this trial are high, yet seemed to be safe and can be considered for use.

In this randomized controlled trial, we aim to evaluate the effect of the combination therapy (vitamin C,thiamine and hydrocortisone) on septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years old or older
* Onset of septic shock within 12 hours

Exclusion Criteria:

* Systemic corticosteroid therapy within the last 3 months before septic shock
* High-dose steroid therapy
* Immunosuppression
* Pregnant
* Known glucose-6 phosphate dehydrogenase (G-6PD) deficiency
* Known hemachromatosis
* Known allergy to vitamin C, hydrocortisone, or thiamine
* Anticipated death from a preexisting disease within 90 days after randomization (as determined by the enrolling physician)
* Refusal of the attending staff or patient family

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
90-day mortality | 90 days after randomization
  Death from any cause at 90 days after the onset of septic shock

SECONDARY OUTCOMES:
ICU mortality | 90 days after randomization
  All-cause mortality at ICU discharge
Hospital mortality | 90 days after randomization
  All-cause mortality at hospital discharge
28-day mortality | 28 days after randomization
  Death from any cause at 28 days after the onset of septic shock

CONTACTS AND LOCATIONS:
Overall Officials: Qingquan Lyu, Master, Principal Investigator — Northern Jiangsu People's Hospital
Locations (1):
- Northern Jiangsu Province people's hospital, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lyu QQ, Zheng RQ, Chen QH, Yu JQ, Shao J, Gu XH. Early administration of hydrocortisone, vitamin C, and thiamine in adult patients with septic shock: a randomized controlled clinical trial. Crit Care. 2022 Sep 28;26(1):295. doi: 10.1186/s13054-022-04175-x. PMID 36171582